CLINICAL TRIAL: NCT01467401
Title: A Multi-National, Multi-Centre, Randomised, Open-Labelled, Parallel Trial Comparing Efficacy and Safety of NovoMix® 30 FlexPen® and Mixtard® 30 Twice Daily Injections in Subjects With Type 2 Diabetes
Brief Title: Efficacy and Safety of NovoMix® 30 in Subjects With Type 2 Diabetes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BIASP-1394
Record Dates: First submitted 2011-11-04; First posted 2011-11-08 (Estimated); Last update posted 2017-02-24 (Actual); Status verified 2017-02

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — insulin aspart, insulin aspart protamine drug combination 30:70; biphasic human insulin 30

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental)
  Interventions: Drug: biphasic insulin aspart
- B (Active Comparator)
  Interventions: Drug: biphasic human insulin

INTERVENTIONS:
Drug: biphasic insulin aspart — Individually adjusted dose. Injected subcutaneously (s.c., under the skin) twice daily
  Arms: A
Drug: biphasic human insulin — Individually adjusted dose. Injected subcutaneously (s.c., under the skin) twice daily
  Arms: B

SUMMARY:
This trial is conducted in Europe. The aim of this trial is to investigate the efficacy and safety of biphasic insulin aspart (NovoMix®30) to that of biphasic human insulin (Mixtard® 30) in subjects with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes for at least 24 months
* Insulin treatment for the pase 3 months
* HbA1c (glycosylated haemoglobin) below 13%
* BMI (Body Mass Index) below 40 kg/m^2
* Ability and willingness to perform self-blood glucose monitoring

Exclusion Criteria:

* Receipt of any investigational drug within 4 weeks prior to this trial
* Treatment of OHAs (Oral Hypoglycaemic Agents) within 4 weeks prior to this trial
* Total daily insulin dosage less than or equal to 1.8 IU/kg

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 292 (Actual)
Dates: Start 2002-08-19 (Actual); Primary Completion 2003-05-15 (Actual); Study Completion 2003-05-15 (Actual)

PRIMARY OUTCOMES:
HbA1c (glycolated haemoglobin)

SECONDARY OUTCOMES:
Prandial increment in blood glucose
7-point blood glucose profile
Number and severity of adverse events
Number and severity of local tolerability issues at the injection site
Number and severity of hypoglycaemic episodes

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (49):
- Denmark (9):
  - Novo Nordisk Investigational Site, Århus C
  - Novo Nordisk Investigational Site, Esbjerg
  - Novo Nordisk Investigational Site, Herning
  - Novo Nordisk Investigational Site, Holbæk
  - Novo Nordisk Investigational Site, Næstved
  - Novo Nordisk Investigational Site, Randers
  - Novo Nordisk Investigational Site, Silkeborg
  - Novo Nordisk Investigational Site, Skive
  - Novo Nordisk Investigational Site, Viborg
- Norway (9):
  - Novo Nordisk Investigational Site, Åsgårdstrand
  - Novo Nordisk Investigational Site, Bekkestua
  - Novo Nordisk Investigational Site, Bergen
  - Novo Nordisk Investigational Site, Haugesund
  - Novo Nordisk Investigational Site, Hønefoss
  - Novo Nordisk Investigational Site, Moelv
  - Novo Nordisk Investigational Site, Oslo
  - Novo Nordisk Investigational Site, Tromsø
  - Novo Nordisk Investigational Site, Vennesla
- Sweden (31):
  - Novo Nordisk Investigational Site, Arvika
  - Novo Nordisk Investigational Site, Avesta
  - Novo Nordisk Investigational Site, Bjuv
  - Novo Nordisk Investigational Site, Broby
  - Novo Nordisk Investigational Site, Färgelanda
  - Novo Nordisk Investigational Site, Gothenburg
  - Novo Nordisk Investigational Site, Grästorp
  - Novo Nordisk Investigational Site, Habo
  - Novo Nordisk Investigational Site, Härnösand
  - Novo Nordisk Investigational Site, Hässleholm
  - Novo Nordisk Investigational Site, Helsingborg
  - Novo Nordisk Investigational Site, Jönköping
  - Novo Nordisk Investigational Site, Karlstad
  - Novo Nordisk Investigational Site, Kristianstad
  - Novo Nordisk Investigational Site, Kristinehamn
  - Novo Nordisk Investigational Site, Kungsbacka
  - Novo Nordisk Investigational Site, Malmo
  - Novo Nordisk Investigational Site, Mellerud
  - Novo Nordisk Investigational Site, Mölndal
  - Novo Nordisk Investigational Site, Norrköping
  - Novo Nordisk Investigational Site, Örebro
  - Novo Nordisk Investigational Site, Östersund
  - Novo Nordisk Investigational Site, Säffle
  - Novo Nordisk Investigational Site, Skövde
  - Novo Nordisk Investigational Site, Stockholm
  - Novo Nordisk Investigational Site, Tomelilla
  - Novo Nordisk Investigational Site, Torsby
  - Novo Nordisk Investigational Site, Trollhättan
  - Novo Nordisk Investigational Site, Tyresö
  - Novo Nordisk Investigational Site, Uddevalla
  - Novo Nordisk Investigational Site, Värnamo

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com